CLINICAL TRIAL: NCT06088888
Title: A Single-arm, Open-label, Dose Escalation + Cohort Expansion Phase 1 Trial on Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of TGRX-678 in Subjects with Refractory or Advanced Chronic Myelogenous Leukemia
Brief Title: TGRX-678 US Phase I for Subjects with Refractory or Advanced Chronic Myelogenous Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen TargetRx, Inc. (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGRX-678-07-101
Record Dates: First submitted 2023-10-08; First posted 2023-10-18 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TGRX-678 (Experimental): Subjects to be treated with the investigational drug TGRX-678
  Interventions: Drug: TGRX-678

INTERVENTIONS:
Drug: TGRX-678 — Participants are given TGRX-678 tablets orally, once daily, at one of the dose levels as pre-determined for the dose escalation sequence or expansion cohorts.

SUMMARY:
The purpose of this single-arm, open-label, dose escalation + cohort expansion study is to evaluate the safety, tolerability, pharmacokinetic and preliminary efficacy of TGRX-678 in Chronic Myelogenous Leukemia patients who had failure with or are intolerant to TKI treatments.

DETAILED DESCRIPTION:
This is the first trial with TGRX-678 conducted to US patients which aims to evaluate the safety profile and preliminary efficacy profile in advanced or refractory CML patients with previous failure or intolerance to TKI treatments. The primary purpose of this study is to evaluate the safety profile of TGRX-678, including determination of the recommended dose for expansion (RDE) and other safety measures of the investigational drug, such as adverse events and abnormal clinical outcomes. Preliminary efficacy profile of TGRX-678 is evaluated based on the changes in peripheral blood cells and disease-associated cytogenetic and molecular markers. Recommended Phase II dose (RP2D) will be determined at end of the study considering safety, tolerability, pharmacokinetic and efficacy data.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study with informed consent;
* At least 18 years of age at the time of screening;
* Any sex;
* Diagnosis of CML-CPduring the screening period;
* Intolerant or resistant to TKI treatments;
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
* Adequate Absolute neutrophil count (ANC), hemoglobin and platelets levels;
* Adequate renal and liver function;
* Normal corrected QT (QTcF) interval as indicated by electrocardiogram (ECG) screening results;
* Negative blood pregnancy test results for female patients of childbearing potential.
* Willing to take highly effective contraceptive measures throughout the trial and for 6 months after last dose of investigational drug for female subjects of child-bearing potential or male subject with female partner of child-bearing potential.

Exclusion Criteria:

* Exposure to other antineoplastic therapies prior to study enrollment;
* Exposure to other investigational agent(s) within 14 days of initiating TGRX-678 therapy;
* Ongoing toxicity from prior therapy greater than grade 1 by CTCAE v. 3 (except alopecia);
* Hematopoietic cell transplantation < 60 days prior to the first dose;
* Evidence of graft versus host disease (GVHD), whether or not requiring immunosuppressive therapy;
* Concomitant immunosuppressive therapy (other than short-term corticosteroid treatment);
* Exposure to drugs related to torsade de pointes;
* Cytological or pathological diagnosis of active central nervous system disorder;
* Significant or uncontrolled cardiovascular diseases as defined in the full clinical protocol;
* Having long QT syndrome, or with family history of idiopathic sudden death or congenital long QT syndrome;
* Uncontrolled hypertension;
* Receipt of Traditional Chinese medication or herbal preparations indicated for anti-cancer purposes within 2 weeks prior to the first dose;
* Severe hemorrhagic disorders unrelated to CML;
* History of pancreatitis;
* History of excessive alcohol use;
* History of elevation in amylase or lipase within 1 year;
* Have Grade 2 or worse interstitial lung disease or interstitial pneumonitis within 4 weeks prior to Screening;
* Uncontrolled hypertriglyceridemia;
* Malabsorption syndrome or other illness that could affect oral absorption.
* Diagnosis of another primary malignancy in the past 3 years;
* Reception of major surgery within 14 days prior to the first dose;
* Active infections that require systemic treatment or other severe infections within 14 days prior to enrollment;
* Known human immunodeficiency virus (HIV) positive; acute or chronic liver disease (including chronic hepatitis B virus (HBV) and hepatitis C virus (HCV) infections);
* Have received or will receive a COVID-19 vaccine within 14 days of study enrollment;
* Have a positive reverse transcriptase polymerase chain reaction (RT-PCR) test result for SARS-CoV-2 within 2 weeks prior to Screening;
* Pregnant or breastfeeding female;
* Female patient of child-bearing potential or male patient who have female partners of child-bearing potential that is unable or unwilling to take highly effective contraceptive measures during the trial and for 6 months after last dose of investigational drug;
* Significant organ dysfunction that could compromise the patient's safety or the evaluation of the drug's safety in the opinion of the investigator or the medical monitor;
* Any condition makes participation in this trial inappropriate in the opinion of the investigator or medical monitor;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Recommended dose for expansion (RDE) | Time Frame: At end of Dose Escalation part of study, an average of 1 year
  To determine the RDE of TGRX-678 in CML patients to be applied in Cohort Expansion part of the study
Safety profile (DLT) | Time Frame: DLT: collect during Cycle 1 (28 days)
  to record and analyse subjects with dose-limiting toxicities (DLTs)
Safety profile (AEs/SAEs) | AE and SAE: through completion of the study, an average of 2 years
  to record and analyse subjects with adverse events (AEs) and serious adverse events (SAEs)
Recommended phase II dose (RP2D) | At completion of the study, an average of 2 years
  To determine the RP2D of TGRX-678 in CML patients for Phase II

SECONDARY OUTCOMES:
Hematologic Response | at screening period, weekly in Cycle 1, bi-weekly in Cycle 2 and monthly starting from Cycle 3 (each cycle is 28 days), an average of 1.5 years
  To record and analyse the hematologic response of subjects. Subjects will be determined whether complete hematologic response (CHR) or no evidence of leukemia (NEL) is reached.
Cytogenetic Response | at screening period, end of every 3 Cycles (each cycle is 28 days), an average of 1.5 years
  To record and analyse the cytogenetic response of subjects subjects will be determined whether partial or complete cytogenetic response (Ph+ < 35%) is reached.
Molecular Response | at screening period, end of every 3 Cycles (each cycle is 28 days), an average of 1.5 years
  To record and analyse the molecular response of subjects Subjects will be determined whether major molecular response (BCR-ABL1 (IS) no more than 0.1%) is reached.
Plasma Cmax | Day 1, 7, 21, 28 of Cycle 1, and Day 28 of Cycle 2, 3 and 5 (each cycle is 28 days)
  Cmax of TGRX-678 as measured in plasma
Plasma Tmax | Day 1, 7, 21, 28 of Cycle 1, and Day 28 of Cycle 2, 3 and 5 (each cycle is 28 days)
  Tmax of TGRX-678 as measured in plasma
Plasma T1/2 | Day 1, 7, 21, 28 of Cycle 1, and Day 28 of Cycle 2, 3 and 5 (each cycle is 28 days)
  T1/2 of TGRX-678 as measured in plasma
Plasma AUClast | Day 1, 7, 21, 28 of Cycle 1, and Day 28 of Cycle 2, 3 and 5 (each cycle is 28 days)
  AUClast of TGRX-678 as measured in plasma
Plasma AUCinf | Day 1, 7, 21, 28 of Cycle 1, and Day 28 of Cycle 2, 3 and 5 (each cycle is 28 days)
  AUCinf of TGRX-678 as measured in plasma
Plasma Cmin | Day 1, 7, 21, 28 of Cycle 1, and Day 28 of Cycle 2, 3 and 5 (each cycle is 28 days)
  Cmin of TGRX-678 as measured in plasma
Plasma AUCss | Day 1, 7, 21, 28 of Cycle 1, and Day 28 of Cycle 2, 3 and 5 (each cycle is 28 days)
  AUCss of TGRX-678 as measured in plasma
Plasma Cmax,ss | Day 1, 7, 21, 28 of Cycle 1, and Day 28 of Cycle 2, 3 and 5 (each cycle is 28 days)
  steady state Cmax of TGRX-678 as measured in plasma
Plasma Tmax,ss | Day 1, 7, 21, 28 of Cycle 1, and Day 28 of Cycle 2, 3 and 5 (each cycle is 28 days)
  steady state Tmax of TGRX-678 as measured in plasma
CL (Clearance) | Day 1, 7, 21, 28 of Cycle 1, and Day 28 of Cycle 2, 3 and 5 (each cycle is 28 days)
  Clearance of TGRX-678 as measured in plasma
Vd (Volume of distribution) | Day 1, 7, 21, 28 of Cycle 1, and Day 28 of Cycle 2, 3 and 5 (each cycle is 28 days)
  Volume of distribution of TGRX-678 as measured in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No